CLINICAL TRIAL: NCT00669136
Title: A Phase I/II Trial Testing Immunization With AFP + GM CSF Plasmid Prime and AFP Adenoviral Vector Boost in Patients With Hepatocellular Carcinoma
Brief Title: Immunization With AFP + GM CSF Plasmid Prime and AFP Adenoviral Vector Boost in Patients With Hepatocellular Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor accrual and limited target patient population for future accrual. Did not complete the Phase 1 portion of the trial.
Sponsor: Lisa H. Butterfield, Ph.D. (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Lisa H. Butterfield, Ph.D., Professor of Medicine, Surgery and Immunology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-101; R01CA104524 (NIH)
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Hepatocellular Carcinoma; Hepatoma; Liver Cancer, Adult; Liver Cell Carcinoma; Liver Cell Carcinoma, Adult; Cancer of Liver; Cancer of the Liver; Cancer, Hepatocellular; Hepatic Cancer; Hepatic Neoplasms; Hepatocellular Cancer; Liver Cancer; Neoplasms, Hepatic; Neoplasms, Liver
Keywords: AFP + GM-CSF Plasmid Prime and AFP Adenoviral Vector Boost; AFP Immunization
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): AFP + GM-CSF Plasmid Prime and AFP Adenoviral Vector Boost
  Interventions: Drug: AFP + GM-CSF Plasmid Prime and AFP Adenoviral Vector Boost

INTERVENTIONS:
Drug: AFP + GM-CSF Plasmid Prime and AFP Adenoviral Vector Boost — AFP + GM-CSF Plasmid Prime and AFP Adenoviral Vector Boost

SUMMARY:
To evaluate the safety, toxicity and immunological effects of adjuvant administration of an experimental therapy consisting on priming with three intramuscular administrations of a plasmid expressing human AFP (phAFP) together with a plasmid expressing human GM-CSF (phGM-CSF), followed by a single intramuscular boost with an AFP adenoviral vector (AdVhAFP) to patients with locoregionally pre-treated hepatocellular carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

Eligible patients must have locoregionally treated HCC and have a prior AFP serum determination over the limit of normality for each laboratory.

* This study will enroll adults over the age of 18.
* Have had HCC with a history of serum AFP determination above the upper limit of normality for each laboratory.
* Both male and female patients may be enrolled. Premenopausal females who have not undergone a surgical sterilization procedure must have a negative pregnancy test prior to treatment. Sexually active females of child-bearing potential are required to use two forms of contraception, including a barrier method, for trial eligibility. Sexually active males should use an appropriate "double barrier" method of birth control (such as female use of a diaphragm, intrauterine device (IUD), or contraceptive sponge, in addition to male use of a condom.
* Be HLA-A2.1 positive (HLA-A*0201) by DNA subtyping, or HLA-A2 positive by flow cytometry with antibodies MA2.1 and BB7.2.
* Stage II to IVa HCC after locoregional therapy (surgical resection, radio-frequency ablation, cryoablation, ethanol injection, chemoembolization and radioembolization).
* Karnofsky Performance Status greater than or equal to 70 percent.
* No evidence of opportunistic infection in the year before enrollment.
* Adequate baseline hematological function as assessed by the following laboratory values within 30 days prior to study entry (day -30 to 0):

Hemoglobin > 9.0 g/dL (patients cannot be transfusion dependent) Platelets > 50,000/mm3 Absolute Neutrophil Count (ANC) > 1,000/mm3

* Conserved liver function with a Child-Pugh Class A or B.
* Ability to give informed consent.

Exclusion Criteria:

Patients who meet any one of the following criteria will be excluded from study entry:

* Any congenital or acquired condition leading to inability to generate an immune response, including concomitant immune suppressive therapy. The ability to adequately respond to recall skin test antigens will be tested before trial entry but a negative response to skin allergens will not be reason for exclusion.
* Concomitant steroid therapy or chemotherapy, or any of these treatments < 30 days before the first vaccination.
* Females of child-bearing potential (premenopausal and not surgically sterilized) must have a negative serum HCG pregnancy test (within Day 14 to Day 0).
* Acute infection: any acute viral, bacterial, or fungal infection, which requires specific therapy excluding HBV or HCV. Acute therapy must have been completed within 14 days prior to study treatment.
* HIV-infected patients (their ability to generate a cellular immune response is altered due to the CD4-dependent immunosuppressive effects of the HIV infection).
* Patients with any underlying conditions which would contraindicate therapy with study treatment (or allergies to reagents used in this study).
* Patients with organ allografts (they require prolonged immunosuppressive therapy).
* Patients with high serum titers of neutralizing anti-adenoviral antibodies (positive at greater than 1:128 dilution by serum AdV blocking assay, expected to be approximately 30% of patients, they have a greatly reduced ability to respond to the AdV boost).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) and Phase II Recommended Dose (P2RD) | 6 months
Immunological response rate in PBMC as indicated by the ELISPOT assay | 6 months

SECONDARY OUTCOMES:
Disease-Free Survival (DFS) | six months
Immunological response rate as indicated by optional DTH | six months
Immunological response rate in PBMC as indicated by the tetramer assay | six months
Immunological response rate in lymph nodes as indicated by the ELISPOT assay | six months

CONTACTS AND LOCATIONS:
Overall Officials: James Pingpank, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of California, Los Angeles, California
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania